CLINICAL TRIAL: NCT01926353
Title: Tissue Bulking Agent -Polyacrylate Polyalcohol Copolymer for Endoscopic Correction of Vesicoureteral Reflux in Children: A Comparative Study
Brief Title: Polyacrylate Polyalcohol Copolymer for Vesicoureteral Reflux
Status: Completed | Type: Observational
Sponsor: St. Luke's Medical Center, Philippines (Other)
Responsible Party: Principal Investigator, Michael E. Chua, Urology Staff, St. Luke's Medical Center, Philippines
Other Study IDs: SLMC13-100
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Vesicoureteral Reflux (VUR); Urinary Tract Infection
Keywords: Vesicoureteral Reflux (VUR); Complicated Urinary Tract Infection; Vantris; Polyacrylate Polyalcohol Copolymer
MeSH Terms: conditions — Vesico-Ureteral Reflux; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Vantris: Patient who categorized as who underwent endoscopic correction procedure, were patients who under general anesthesia performed by a single experienced surgeon using a 10Fr Storz® cystoscope with PPC (Vantris®) subureteral or intraureteral injection, or a combination of both techniques, depending on the anatomy of the ureteral meatus and VUR grade.
- Cohen reimplantation: Patient underwent surgical management were all had ureteral re-implatation with Cohen technique done by single experienced pediatric urologist.
- Continuous Antibiotic Prophylaxis: Group of patient treated with conservative management were children treated with culture guided antibiotics and maintained on 1st or 2nd generation cephalosporin as continuous antibiotic prophylaxis until time of 1 year follow-up.

SUMMARY:
Endoscopic correction of VUR has gained its popularity due to its less invasiveness, associated low morbidity and short hospital stay. Although short term follow-up had justified their efficacy; however, long term recurrence and complications following endoscopic correction were also being reported in the literatures (6). Currently, there are insufficient evidences on the efficacy and safety of biocompatible tissue augmenting materials used for endoscopic correction of VUR; particularly on the new tissue bulking agents. (6) Polyacrylate polyalcohol copolymer (PPC)-Vantris ® (Promedon, Cordoba, Argentina) is the newest tissue augmenting biocompatible Acrylics used for endoscopic correction of VUR.

ELIGIBILITY:
Inclusion Criteria:

* Included patients for the study were only those who had 1- 3months and >1year post-treatment follow-up study with voiding cystourethrogram (VCUG), kidney ultrasound, dimercaptosuccinic acid(DMSA) renal scan, and urine culture.

Exclusion Criteria:

* Excluded cases were patients who had VUR grade 1 and grade 5, no complete follow-up work ups, concomitant neurogenic bladder, anatomical malformation of the urinary tract (obstruction, complete duplicated pelvocaliceal system), previous surgical or endoscopic procedures, and suspected or confirmed dysfunctional voiding by clinical findings or abnormal results (irregular bladder wall, diverticulum) on VCUG or urodynamic study.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children diagnosed with primary VUR grade 2-4 from 2006-2012 treated by a single urologist with different treatment modalities- conservative continuous antibiotic prophylaxis, endoscopic correction with PPC and open ureteral re-implantation with Cohen technique.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rate of Treatment success | 3 months, 1 year
  Rate of complete resolution of VUR on follow-up VCUG at 3 months and 1 year.

SECONDARY OUTCOMES:
Rate of renal scar development | at 3 months, 1 year
  The rate of Renal scarring is defined as consistent decreased tracer activity noted in follow-up DMSA scan.
Length of VUR treatment related hospital stay | 1 year
  Number of hospital days incurred related to VUR treatment, such as hospital admission on treatment period, recovery period, and subsequent admissions for complicated UTI secondary to VUR.
Rate of failed treatment response | 3 months, 1 year
  Rate of VUR with resoultion noted on 3 month follow-up; however, VUR noted on 1 year VCUG follow-up. Failed treatment defined as persistent VUR or VUR grade progressed despite treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelino L Morales, MD, Study Director — Institute of Urology, St. Luke's Medical Center, Quezon City, Philippines
Locations (1):
- St. Luke's Medical Center, Quezon City, NCR, Philippines